CLINICAL TRIAL: NCT06223516
Title: A Multicenter, Phase 1b, Open-label Study of Etentamig (ABBV-383) Administered Subcutaneously in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of ABBV-383 Assessing Adverse Events and Clinical Activity With Subcutaneous (SC) Injection in Adult Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-001; 2023-507901-32-00 (Other: EU CT)
Record Dates: First submitted 2024-01-17; First posted 2024-01-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; ABBV-383; Etentamig
MeSH Terms: conditions — Multiple Myeloma | interventions — Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Etentamig Dose A (Experimental): Participants will receive Dose A of Etentamig as a subcutaneous (SC) injection and intravenous (IV) infusions, during the 151 week study duration.
  Interventions: Drug: Subcutaneous (SC) Etentamig; Drug: Intravenous (IV) Etentamig
- Etentamig Dose B (Experimental): Participants will receive Dose B of Etentamig as an SC injection and IV infusions, during the 151 week study duration.
  Interventions: Drug: Subcutaneous (SC) Etentamig; Drug: Intravenous (IV) Etentamig
- Etentamig Expansion (Experimental): Participants will receive the selected dose from Arm A of Etentamig as SC injections, during the 151 week study duration.
  Interventions: Drug: Subcutaneous (SC) Etentamig

INTERVENTIONS:
Drug: Subcutaneous (SC) Etentamig — SC Injection
Drug: Intravenous (IV) Etentamig — IV Infusion
  Arms: Etentamig Dose A; Etentamig Dose B

SUMMARY:
Multiple myeloma (MM) is a cancer of the blood's plasma cells. The cancer is typically found in the bones and bone marrow (the spongy tissue inside of the bones) and can cause bone pain, fractures, infections, weaker bones, and kidney failure. Treatments are available, but MM can come back (relapsed) or may not get better (refractory) with treatment. This is a study to determine the safety and pharmacokinetics of Etentamig (ABBV-383) in adult participants with relapsed/refractory (R/R) MM.

Etentamig (ABBV-383) is an investigational drug being developed for the treatment of R/R MM. This study is broken into 3 Arms: Arm A with 2 parts and Arm B as an expansion. Participants will receive ABBV-383 as a subcutaneous (SC) injection and intravenous (IV) infusion in Arm A and SC injections of ABBV-383 in Arm B. Around 55 adult participants with relapsed/refractory multiple myeloma will be enrolled at approximately 15 sites across the world

In Arm A participants will receive one of two doses of Etentamig (ABBV-383) as an SC injection and (IV) infusions, during the 151 week study duration. In Arm B, participants will receive the selected dose from Arm A as SC injections, during the 151 week study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance of <= 2.
* Participants with relapsed or refractory multiple myeloma who have received 3-5 prior lines of therapies and with prior triple class exposure including a proteasome inhibitor, anti-CD38 monoclonal antibody and an immunomodulatory drug.
* Must be naïve to treatment with ABBV-383.

Exclusion Criteria:

- Received B-cell maturation antigen (BCMA)xCD3 bispecific antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Cytokine Release Syndrome (CRS) Events | Up to 2 cycles (56 days)
  Cytokine Release Syndrome events will be graded using American Society for Transplantation and Cellular Therapy (ASTCT), with a higher grade indicating higher severity.
Percentage of Participants Experiencing Immune Cell-Associated Neurotoxicity Syndrome (ICANS) Events | Up to 2 cycles (56 days)
  ICANS events will be graded using ASTCT, with a higher grade indicating higher severity.
Maximum Observed Concentration (Cmax) of ABBV-383 | Up to 32 weeks
  Cmax of ABBV-383.
Time to Cmax (Tmax) of ABBV-383 | Up to 32 weeks
  Tmax of ABBV-383.
Trough Concentration (Ctrough) of ABBV-383 | Up to 32 weeks
  Ctrough of ABBV-383.
Area Under the Plasma Concentration-time Curve (AUC) of ABBV-383 | Up to 24 weeks
  AUC of ABBV-383.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  The ORR is defined as the percentage of participants who achieve a best overall response of confirmed PR or better determined by international myeloma working group (IMWG) criteria, prior to the initiation of subsequent myeloma therapy.
Percentage of Participants Achieving Stringent Complete Response (sCR), | Up to 24 months
  sCR is defined as participants achieving negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, < 5% plasma cells in bone marrow, normal free light chain (FLC) ratio, and Absence of clonal cells in bone marrow by immunohistochemistry.
Percentage of Participants Achieving Complete Response (CR) | Up to 24 months
  CR is defined as participants achieving negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, < 5% plasma cells in bone marrow, and for participants in whom the only measurable disease is by serum FLC levels, a normal FLC ratio.
Percentage of Participants Achieving Very Good Partial Response (VGPR) | Up to 24 months
  VGPR is defined as participants achieving serum and urine M-protein detectable by immunofixation but not on electrophoresis, >= 90% reduction in serum M-protein plus urine, and for participants in whom the only measurable disease is by serum FLC levels, >= 90% decrease in the difference between involved and uninvolved FLC levels.
Percentage of Participants Achieving Partial Response (PR) | Up to 24 months
  PR is defined as participants achieving >= 50% reduction of serum M-protein, reduction in 24-hour urinary M-protein by >= 90% as noted in the protocol, >= 50% reduction in the size of soft tissue plasmacytomas is also required, if present at baseline.
Duration of Response (DoR) | Up to 24 months
  DoR will be defined as the time from the date of first response [partial response (PR) + VGPR + complete response (CR) + stringent complete response (sCR)] to the earliest occurrence of progressive disease, or death, whatever occurs first.
Progression Free Survival (PFS) | Up to 24 months
  PFS is defined as the duration from the date of randomization to the date of confirmed disease progression (PD) per international myeloma working group (IMWG) criteria, or death, whichever occurs first.
Time to Response (TTR) | Up to 24 months
  TTR is defined as the number of months from the date of first dose to the date of best overall response of CR or PR ('responders') determined by IMWG criteria.
Immunogenicity of ABBV-383 as Determined by Anti-Drug Antibodies (ADAs) | Up to 27 months
  Incidence and concentration of ADAs.
Immunogenicity of ABBV-383 as Determined by Neutralizing Anti-Drug Antibodies (NAbs) | Up to 27 months
  Incidence and concentration of NAbs.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United States (7):
  - Mayo Clinic Arizona /ID# 260799, Phoenix, Arizona
  - Mayo Clinic Hospital Jacksonville /ID# 262808, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center /ID# 260798, Miami, Florida
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 261050, Ann Arbor, Michigan
  - Mayo Clinic - Rochester /ID# 262807, Rochester, Minnesota
  - Atrium Health Wake Forest Baptist Medical Center /ID# 260807, Winston-Salem, North Carolina
  - Wisconsin Medical Center /ID# 261085, Milwaukee, Wisconsin
- Germany (3):
  - Universitaetsklinikum Frankfurt /ID# 260442, Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln /ID# 260445, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 260444, Hamburg
- Israel (3):
  - Hadassah Medical Center-Hebrew University /ID# 261446, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 261699, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 261525, Tel Aviv, Tel Aviv
- Japan (2):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital /ID# 265286, Nagoya, Aichi-ken
  - Kindai University Hospital /ID# 266016, Sakai-shi, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-001